CLINICAL TRIAL: NCT03193905
Title: Preventing Inadvertent Hypothermia in Patients Undergoing Major Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mia Nørgaard Granum, Anaesthetic nurse, Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BFAU blanket 2016
Record Dates: First submitted 2017-01-11; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-01

CONDITIONS: Hypothermia Following Anesthesia; Neurosurgery; Scoliosis; Kyphosis; Forced Air Warming; Major Spinal Fusion
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cotton blanket (Other): 30 hypothermia patients undergo the standard procedure with a cotton blanket during major spinal surgery
  Interventions: Procedure: Cotton blanket - control group
- Bairhugger Full Access Underbody blanket (Other): 30 hypothermia patients undergo the Bairhugger Full Access Underbody blanket procedure during major spinal surgery (new procedure)
  Interventions: Procedure: Bairhugger Full Access Underbody Blanket

INTERVENTIONS:
Procedure: Bairhugger Full Access Underbody Blanket — 30 patients undergo new procedure with a Bairhugger Full Access Underbody Blanket
  Arms: Bairhugger Full Access Underbody blanket
Procedure: Cotton blanket - control group — 30 patients undergo standard procedure with a cotton blanket
  Arms: Cotton blanket

SUMMARY:
Background

Major spinal surgery tend to be lengthy with an increased risk of hypothermia. A quality improvement project of patients undergoing major spinal surgery showed that 67 % were hypothermic at the beginning of surgery. Several patients expressed a feeling of coldness at the arrival of the operating theatre.

Aim

To evaluate if Bairhuggers Full Access Underbody blanket can prevent hypothermia at initiation if used as prewarming and intraoperative warming compared to the results from the local quality improvement project. In addition we aim to explore patients´ experiences of comfort in relation to their temperature.

Method

Temperature of patients undergoing major spinal surgery (n=30) will be assessed at arrival to the theatre, after insertion of bladder catheter, at the start and end of surgery using a bladder temperature. The patients´ experiences of comfort will be evaluated with a 5 point Likert at the arrival to the operating theatre and after ten minutes of active prewarming with Bairhuggers Full Access Underbody blanket. Preoperatively ten randomly chosen patients will be observed and later interviewed in order to obtain further information regarding their experiences of comfort in relation to their temperature.

Conclusion and perspectives

By increasing the investigators knowledge on Bairhuggers Full Access Underbody blanket and its effects in preventing hypothermia as well as gaining insight to patients´ experiences of comfort in relation to temperature, the investigators anticipate to improve pre-anesthetic care and minimize risk factors associated with hypothermia for patients undergoing major spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective major spinal surgery
* Patients ≥ 14 years
* Danish language

Exclusion Criteria:

* Patients> 110 kg
* Patients with a temperature > 37.5 ° C
* Patients with a temperature ≤ 35 ° C
* Cognitive impairment to such an extent that the patient does not understand the purpose of, nor is able to cooperate, with the project

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Core temperature > 36 degrees Celsius | Althrough completion of the study 5 months from now
  Core temperature at the start of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mia Nørgaard Granum, Principal Investigator — Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: No